CLINICAL TRIAL: NCT05964998
Title: Investigating Non-invasive Brain Stimulation to Enhance CBT in Intensive Treatment-seeking Patients With OCD
Brief Title: Pilot Study of CBT With tDCS for Adults Being Treated for Obsessive Compulsive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find patients willing to consent; declined for various reasoning: e.g., time commitment for the study, concerns about electrode gel in the hair, and concerns about potentially being randomized to a control group.
Sponsor: Rogers Behavioral Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-ROGE-103
Record Dates: First submitted 2023-04-03; First posted 2023-07-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; transcranial direct current stimulation; tDCS; Cognitive Behavior Therapy; CBT
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants randomized to either active tDCS stimulation or sham.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active stimulation (Experimental)
  Interventions: Device: transcranial direct current stimulation
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Current will increase to 1.5 milliamps within 30 seconds and then maintain for 20 minutes
  Arms: Active stimulation
Device: Sham transcranial direct current stimulation — Current will increase up to 1.5 milliamps within 30 seconds and then decrease back down over the next 30 seconds to 0 milliamps; subjects will received 0 milliamps for 20 minutes
  Arms: Sham stimulation

SUMMARY:
This pilot study aims to compare the effect of transcranial direct current stimulation (tDCS) versus sham stimulation, delivered immediately prior to cognitive-behavioral therapy (CBT) for obsessive-compulsive disorder (OCD), on patient-reported outcomes. The investigator hypothesize that patients who receive active stimulation will experience greater improvement in OCD symptoms than those who receive sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Obsessive-Compulsive Disorder (OCD)
* Resident of state of Wisconsin
* Enrolled in OCD Intensive Outpatient Program (IOP) at Rogers Behavioral Health in Oconomowoc, WI
* Ability to communicate effectively using written and spoken English

Exclusion Criteria:

* Metal in the body of any kind (e.g., braces, pacemakers, metal plates or screws, intracranial electrodes, implanted devices/defibrillators, prostheses)
* Currently taking medication that reduces seizure threshold (e.g., clomipramine)
* Cranial pathologies (e.g., holes, plates)
* History of seizure or black-out concussion
* Pregnancy
* Previous treatment at Rogers Behavioral Health

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale - Self-Report from admission to discharge | Up to 12 weeks
Change in Quick Inventory of Depressive Symptomology from admission to discharge | Up to 12 weeks

SECONDARY OUTCOMES:
Number of treatment days between admission and discharge | Up to 12 weeks
Change in Obsessive-Compulsive Inventory-Revised from admission to discharge | Up to 12 weeks
Change in Quality of life enjoyment and satisfaction questionnaire - short form from admission to discharge | Up to 12 weeks
Change in Intolerance of uncertainty scale from admission to discharge | Up to 12 weeks
Change in Subjective units of distress from admission to discharge | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C Riemann, PhD, Principal Investigator — Rogers Behavioral Health
Locations (1):
- Rogers Behavioral Health, Oconomowoc, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No